CLINICAL TRIAL: NCT02269436
Title: A Multi-centre, Open-label, follow-on Study to Assess Long-term Safety and Tolerability of Intracerebroventricular Administration of sNN0029 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: A follow-on Study to Assess Long-term Safety and Tolerability of i.c.v Administration of sNN0029 in Patients With ALS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues with development and supply of infusion system for delivery of IMP. Lack of favorable benefit risk ratio in sNN0029-003 study (review of interim data).
Sponsor: Newron Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sNN0029-004; 2012-005034-11 (EudraCT Number)
Record Dates: First submitted 2014-10-08; First posted 2014-10-21 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sNN0029 infusion solution (Experimental)
  Interventions: Drug: sNN0029 infusion solution

INTERVENTIONS:
Drug: sNN0029 infusion solution — 4 µg/day, continuous i.c.v administration

SUMMARY:
This is an open-label, follow-on phase 1 study to assess the long-term safety and tolerability of continuous i.c.v administration of 4 μg sNN0029/day in patients with ALS who previously participated in study sNN0029-003

DETAILED DESCRIPTION:
This is an open-label, follow-on phase 1 study to assess the long-term safety and tolerability of continuous i.c.v administration of sNN0029 infusion solution in patients with ALS.

Eighteen patients who previously participated in study sNN0029-003 will receive continuous administration of 4 μg sNN0029/day via i.c.v. infusion with the Medtronic SynchroMed® II Infusion System. The sNN0029 infusion solution is intended to be an add-on treatment to other treatments for ALS.

The assessments performed at the last visit in study sNN0029-003 will serve as the baseline values for patients included in study sNN0029-004 and be the start of sNN0029 treatment for all patients (Study Day 1; Visit 1). In order to not reveal the blind in study sNN0029-003, the patients will return to hospital on Day 3 and stay to Day 6 (Visit 2). During these days, the sNN0029 begins to exit the i.c.v. catheter tip in the ventricle of the brain.

Patients will return to the hospital on Day 11 (Visit 3) for a refill of sNN0029 and adjustment of the infusion pump flow rate. After this, the patient will return to the clinic on Day 39 (Visit 4) for a sNN0029-refill of infusion pump and assessments. Thereafter the patients will visit the hospital on a monthly basis (every 28 days ± 2) to perform refills and make assessments every 3 months.

Treatment in study sNN0029-004 may continue unless safety concerns warrant discontinuation of therapy, until patients choose to withdraw from the study, experience treatment related toxicity or intolerance, are deemed to be unsuitable to continue treatment by the investigator, or die

ELIGIBILITY:
Inclusion Criteria:

1. Previous participation in sNN0029-003 with completion of 12 weeks study without clinically significant safety concerns
2. Intact continuity of the Medtronic SynchroMed® II Infusion System as judged by X-ray of head and abdominal area
3. Clinical diagnosis of ALS classified as definite, or probable with or without additional laboratory evidence, according to the revised WFN El Escorial criteria
4. Patient has been given written and verbal information about the continuation study, has had the opportunity to ask questions about the study, and understands the time and procedural commitments
5. Patient has given oral and / or signed consent (written) to participate in the study. In the event that a patient who gives oral informed consent is not physically able to sign the informed consent form (ICF) due to disease progression, a witness may sign the informed consent form on the patient's behalf

Exclusion Criteria:

1. Hypertension defined as blood pressure >160 mmHg systolic or >90 mmHg diastolic
2. Ophthalmological examination (fundus photography, visual acuity and perimetry) with any clinically significant findings that imply safety concerns for this study.
3. Diagnosis of diabetes mellitus
4. Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that cannot be not managed optimally due to:

   * Anatomical factors at or near the implant site (e.g., vascular abnormalities, neoplasms, or other abnormalities)
   * Underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., haemophilia, Von Willebrand's disease, liver disease, or other medical conditions)
5. Presence of additional risk factors for thromboembolism such as obesity (Body mass index [BMI] > 35) or use of oestrogens including combined contraceptive pills
6. Clinically significant abnormalities in haematology or clinical chemistry parameters as assessed by the investigator
7. Ongoing medical condition that according to the investigator would interfere with the conduct and assessments in the study. Examples are medical disability (e.g., severe degenerative arthritis, compromised nutritional state, peripheral neuropathy) that would interfere with the assessment of safety and efficacy of investigational product or device performance, or would compromise the ability of the patient to undergo study procedures (e.g., MRI), or to give informed consent
8. For women only: pregnant, breast feeding and/or for fecund women unwillingness to use adequate contraception during the trial such as:

   * Established use of oral, injected or implanted hormonal methods of contraception that do NOT contain oestrogens
   * Placement of an intrauterine device
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number Patients with Adverse Events as a measure of Safety and Tolerability | At 24 Months
  Number of patients with events will be analysed primarily at 24 months of study duration. The study may be extended on a 6-monthly basis for as long as there are patients that tolerate, and are still eligible to receive, the study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Philip Van Damme, Leuven, Belgium
- Leonard van den Berg, Utrecht, Netherlands